CLINICAL TRIAL: NCT02786810
Title: Contrast Enhanced Ultrasound for Evaluation of Reflux Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1504311FB
Record Dates: First submitted 2016-05-17; First posted 2016-06-01 (Estimated); Results first posted 2018-04-04 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2016-05

CONDITIONS: Urinary Tract Infection; Vesicoureteral Reflux
MeSH Terms: conditions — Urinary Tract Infections; Vesico-Ureteral Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast (Other): All subjects will be recruited into this arm. All subjects will receive 0.03 ml/kg IV sulfur hexafluoride type-a lipid microspheres one time, unless a second, adjusted dose is necessary.
  Interventions: Drug: Sulfur hexafluoride type-a lipid microspheres

INTERVENTIONS:
Drug: Sulfur hexafluoride type-a lipid microspheres — Used as a contrast to enhance renal ultrasound
  Other Names: Lumason®

SUMMARY:
The study will be evaluating the efficacy and safety of a contrast drug in pediatric renal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age more than or equal to 8 years
* Patient with history of urinary tract infection (UTI) and history of Voiding Cystourethrogram (VCUG) for vesicoureteral reflux
* Candidate for Dimercaptosuccinic acid (DMSA) scan or scan for renal scar
* Demonstration of renal scarring by DMSA scan or renal ultrasound without contrast

Includes healthy volunteers

Exclusion Criteria:

* Age less than 8years
* Allergy to contrast or related products
* Cardiac shunt/ congenital heart anomalies
* Abnormal baseline ECG
* Open heart surgery
* Evidence of retinopathy
* Patient in intensive care
* Unable to comply with study requirement
* History of emphysema
* Unable to maintain oxygen saturation of 92% on at room air
* Pregnancy and lactation

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hains, M.D., Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrast
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Contrast
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Visualization of Renal Scars Compared to Previous Imaging
Description: The study will evaluate the contrast agent's ability to enable the ultrasound to produce adequate images of the kidneys as compared to the subject's previous renal imaging. This outcome will be measured in percentage of scars visualized by other imaging methods that were detected by using the contrast agent.
Time Frame: 1 hour
Population: In addition to the 7 patients analyzed, 3 participants were excluded from this analysis because they did not have previous scars to analyze.
Measure: Number; unit: Percentage of previous scars visualized
Arm/Group | Contrast
Number analyzed (Participants) | 7
Percentage of previous scars visualized | 100

2. Secondary Outcome: Number of Participants With Adverse Events Related to the Study Drug.
Description: The study will evaluate how many people experience adverse events, specifically the two most common effects (headache and nausea), during the study or during the week following the study.
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Contrast
Number analyzed (Participants) | 10
participants | 1

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Contrast
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contrast (N=10)
Mild Headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No